CLINICAL TRIAL: NCT00003994
Title: Intergroup Protocol for Treatment of Children With Hepatoblastoma
Brief Title: Combination Chemotherapy With or Without Amifostine in Treating Young Patients With Liver Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P9645; NCI-2012-02306 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-P9645 (Other: Children's Oncology Group); CCG-P9645 (Other: Children's Cancer Group); POG-9645 (Other: Pediatric Oncology Group); CDR0000067200 (Other: Clinical Trials.gov); U10CA098543 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Childhood Hepatoblastoma; Recurrent Childhood Liver Cancer; Stage I Childhood Liver Cancer
MeSH Terms: conditions — Hepatoblastoma | interventions — Cisplatin; Vincristine; Fluorouracil; Amifostine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (cisplatin, vincristine sulfate, fluorouracil) (Experimental): Patients receive therapeutic conventional surgery (tumor resection). Patients receive cisplatin IV over 4 hours on day 1, vincristine sulfate IV on days 3, 10, and 17, and fluorouracil on day 3.
  Interventions: Procedure: therapeutic conventional surgery; Drug: cisplatin; Drug: vincristine sulfate; Drug: fluorouracil
- Arm II (cisplatin, vincristine, fluorouracil, amifostine) (Experimental): Patients receive therapeutic conventional surgery (tumor resection). Patients receive treatment as in arm I with the addition of amifostine trihydrate IV over 15 minutes prior to cisplatin on day 1.
  Interventions: Procedure: therapeutic conventional surgery; Drug: cisplatin; Drug: vincristine sulfate; Drug: fluorouracil; Drug: amifostine trihydrate
- Arm III (carboplatin, cisplatin) (Experimental): Patients receive therapeutic conventional surgery (tumor resection). Patients receive carboplatin IV over 1 hour on day 1 and cisplatin IV over 4 hours on day 15.
  Interventions: Procedure: therapeutic conventional surgery; Drug: cisplatin; Drug: carboplatin
- Arm IV (carboplain, cisplatin, amifostine) (Experimental): Patients receive therapeutic conventional surgery (tumor resection). Patients receive treatment as in arm III with the addition of amifostine trihydrate IV over 15 minutes prior to carboplatin on day 1.
  Interventions: Procedure: therapeutic conventional surgery; Drug: cisplatin; Drug: amifostine trihydrate; Drug: carboplatin

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Undergo surgical resection
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
  Arms: Arm I (cisplatin, vincristine sulfate, fluorouracil); Arm II (cisplatin, vincristine, fluorouracil, amifostine)
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
  Arms: Arm I (cisplatin, vincristine sulfate, fluorouracil); Arm II (cisplatin, vincristine, fluorouracil, amifostine)
Drug: amifostine trihydrate — Given IV
  Other Names: ethiofos; Ethyol; gammaphos; WR-2721
  Arms: Arm II (cisplatin, vincristine, fluorouracil, amifostine); Arm IV (carboplain, cisplatin, amifostine)
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
  Arms: Arm III (carboplatin, cisplatin); Arm IV (carboplain, cisplatin, amifostine)

SUMMARY:
Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy. It is not yet known which chemotherapy regimen is most effective for children and young adults with liver cancer. This randomized phase III trial is studying giving combination chemotherapy together with amifostine to see how well it works compared to combination chemotherapy alone in treating patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the response and efficacy of amifostine (amifostine trihydrate) in reducing the toxicity associated with platinum agents.

II. To test whether there is any effect of amifostine on event-free survival by comparing outcome of those treated with amifostine to those treated without on this study and with historic controls.

SECONDARY OBJECTIVES:

I. To estimate the event-free survival of patients with stage I pure fetal histology treated with surgery alone.

II. To estimate the efficacy of amifostine in reducing the toxicity associated with cisplatinum in children with resected tumors receiving treatment 01 by randomizing to receive or not receive amifostine.

III. To collect tumor tissue in all patients for cytogenetic and genetic analysis in order to prospectively analyze biologic features and prognosis of patients with detailed treatment history, and to provide a resource for future biologic studies in hepatoblastoma.

IV. To assess the prognostic significance with respect to event-free survival of hepatoblastoma pathologic variants in patients with stage I tumors treated with surgery and chemotherapy (cisplatin + 5FU + vincristine).

OUTLINE: This is a randomized study. Patients are stratified according to disease stage (stage I pure fetal histology vs stage I other histology or stage II [stage II closed to accrual as of 11-25-03] vs stage III or IV [stages III and IV closed to accrual as of 11-25-03]). Patients are randomized to one of four treatment arms. (Arms III and IV closed to accrual as of 4-5-02) (Arm II closed to accrual as of 11-25-03)

All patients undergo surgical resection or attempted resection of tumor. Patients with pure fetal histology achieving complete tumor resection receive no further treatment. All other patients receive postoperative chemotherapy.

Arm I: Patients receive cisplatin IV over 4 hours on day 1, vincristine IV on days 3, 10, and 17, and fluorouracil on day 3.

Arm II (closed to accrual as of 11-25-03): Patients receive treatment as in arm I with the addition of amifostine IV over 15 minutes prior to cisplatin on day 1.

Arm III (closed to accrual as of 4-5-02): Patients receive carboplatin IV over 1 hour on day 1 and cisplatin IV over 4 hours on day 15.

Arm IV (closed to accrual as of 4-5-02): Patients receive treatment as in arm III with the addition of amifostine IV over 15 minutes prior to carboplatin on day 1.

Treatment repeats every 3 weeks for 4 courses in arms I and II (arm II closed to accrual as of 11-25-03) and every 4 weeks for 4 courses in arms III and IV (arms III and IV closed to accrual as of 4-5-02) in the absence of disease progression or unacceptable toxicity. Patients with stage III or IV disease (stages III and IV closed to accrual as of 11-25-03) undergo second look surgery and receive 2 additional courses of chemotherapy if achieving complete response after surgery.

Patients are followed monthly for 6 months, every 2 months for 2 years, every 3 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 356 patients will be accrued for this study within 5.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven hepatoblastoma

  * Any stage allowed(stages II-IV closed to accrual as of 11-25-03)
* Stratum 1 (stage I):

  * Pure fetal histology
  * Complete surgical resection of tumor
* Stratum 2 (stages I or II) (stage II closed to accrual as of 11-25-03), meeting 1 of the following criteria:

  * Complete resection of tumor with histology other than pure fetal
  * Gross resection of tumor, including resected tumors with preoperative/intraoperative rupture
* Stratum 3 (stages III or IV) (stages III and IV closed to accrual as of 11-25-03), meeting 1 of the following criteria:

  * Unresectable tumors

    * Partial resection of tumor with measurable residual disease OR lymph node involvement
  * Measurable metastatic disease to lungs or other organs
* No hepatocellular carcinoma
* Creatinine normal for age
* Glomerular filtration rate normal for age
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior biologic therapy
* No prior chemotherapy
* No prior endocrine therapy
* No prior radiotherapy
* See Disease Characteristics
* No prior therapy except tumor resection

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 277 (Actual)
Dates: Start 1999-03; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) rates | Up to 8 years
  EFS rates will be estimated using the method of Kaplan and Meier. Survival curves will be compared using stratified logrank tests.
Toxicity rates assessed using National Cancer Institute (NCI) Common Toxicity Criteria (CTC) | Up to 8 years
  For comparing the toxicity rates in the +/- amifostine arms, stratified binomial test for proportions (Mantel-Haenszel) will be used assuming no qualitative interaction between the two chemotherapy regimens and amifostine trihydrate.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Katzenstein, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States